CLINICAL TRIAL: NCT01679561
Title: Phase 4 Study of the Efficacy of Intralipid Treatment in Patients With Recurrent Implantation Failure and Miscarriages With High Peripheral and Uterine Natural Killer Cells
Brief Title: Intralipid Therapy for Recurrent Implantation Failure and Recurrent Miscarriages: Is it a Hope or Myth?A Randomized Clinical Trial
Acronym: ILRIFRM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, M D, Woman's Health University Hospital, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILRIFRM
Record Dates: First submitted 2012-08-20; First posted 2012-09-06 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy Complicated by Low Implantation
Keywords: implantation failure; recurrent abortion; intralipid
MeSH Terms: conditions — Abortion, Habitual | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intralipids (Experimental): Two hundreds patients (group1) with abnormal NK activity results (NKa)will receive intralipids 20% i.v. (9 mg/mL total blood volume -corresponds to 2 mL of intralipids 20% diluted in 250 mL saline; or 18 mg/mL - corresponds to 4 mL of intralipids 20% diluted in 250 mL saline) infusions and their NKa will be tested periodically. The determination of NK cell function will be performed by flow cytometry using K562 cells as targets,then follow up of the patients by the Doppler of endometrial blood follow at the time of luteal phase,and the clinical pregnancy rate.Group(2)of 180 patients will receive placebo.
  Interventions: Drug: intralipid

INTERVENTIONS:
Drug: intralipid — intravenous intralipid 20% is given to the patients known to be have either recurrent failed IVF, RPL

SUMMARY:
Both organ-specific and systemic autoimmunity are associated with an increased prevalence of recurrent miscarriage and reproductive failure, rendering the role of the maternal immunological system in fertility a key concept. It is believed by some that central to this theme is the maternal cytokine profile, with particularly T-helper (Th) cells. Immune modulating therapies have therefore been mooted as potential therapeutic strategies. Recent reports of high pregnancy rates achievable in women with RIF have added fuel to the debate regarding the effectiveness of intralipids in modulating the immune system.

DETAILED DESCRIPTION:
The investigators would like to assess if that intralipids therapy is an effective treatment for women undergoing repeated failed assisted reproduction cycles and recurrent miscarriages against traditional methods in randomised clinical trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent unexplained failed IVF, ICSI.
2. Recurrent unexplained miscarriages.
3. High level of peripheral and uterine NK.

Exclusion Criteria:

1. Age above forty years old.
2. Antiphospholipid syndrome (lupus anticoagulant and/or anticardiolipin antibodies [IgG or IgM]); other recognised thrombophilic conditions (testing according to usual clinic practice).
3. Intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram, or hysteroscopy).
4. Fibroids distorting uterine cavity.
5. Abnormal parental karyotype.
6. Other identifiable causes of recurrent miscarriages (tests initiated only if clinically indicated) e.g., diabetes, thyroid disease and systemic lupus erythematosus (SLE).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of intralipid on normalization of nk level and rate of clinical pregnancy . | 2 ys
  Two hundreds patients (group1) with abnormal NK activity results (NKa)will receive intralipids 20% i.v. (9 mg/mL total blood volume -corresponds to 2 mL of intralipids 20% diluted in 250 mL saline; or 18 mg/mL - corresponds to 4 mL of intralipid 20% diluted in 250 mL saline) infusions and their NKa will be tested periodically. The determination of NK cell function will be performed by flow cytometry using K562 cells as targets,then follow up of the patients by the Doppler of endometrial blood follow at the time of luteal phase,and the clinical pregnancy rate.Group(2)of 200 patients will receive other routine measures.

SECONDARY OUTCOMES:
the rate of continuation of pregnancy beyond 12 weeks of pregnancy,the adverse effects related to the drug. | 2 ys
  Two hundreds patients (group1) with abnormal NK activity results (NKa) will receive intralipids 20% i.v. (9 mg/mL total blood volume -corresponds to 2 mL of intralipid 20% diluted in 250 mL saline; or 18 mg/mL - corresponds to 4 mL of intralipid 20% diluted in 250 mL saline) infusions and their NKa were tested periodically. The determination of NK cell function will be performed by flow cytometry using K562 cells as targets,then follow up of the patients by the Doppler of endometrial blood follow at the time of luteal phase,and the clinical pregnancy rate.Group(2)of 200 patients will receive routine measures.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, M D, Principal Investigator — Faculty of medicine,Assiut university,Egypt
Locations (1):
- Women's Health Hospital, Asyut, Egypt